CLINICAL TRIAL: NCT04716764
Title: Evaluation of The Relationship Between Dietary Advanced Glycation End Products With Inflammation and Oxidative Stress in Breast Cancer Patients
Brief Title: Dietary Advanced Glycation End Products, Inflammation and Oxidative Stress in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Hacettepe University (Other); Turkish Society of Medical Oncology (Unknown)
Responsible Party: Principal Investigator, Şenay Burçin Alkan, Lecturer, Necmettin Erbakan University
Other Study IDs: dAGEs
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Female
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Residual serum samples taken from participants will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: The study will include female individuals aged 19-64 years who applied to Necmettin Erbakan University Meram Medical Faculty General Surgery and Medical Oncology Departments and were diagnosed with breast cancer for the first time and volunteering to participate in the study. Patients with breast cancer will be followed up before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy.
  Interventions: Other: 3-Day Food Intake Record
- Healthy (Control) participants: The control group consists of healthy adult women who applied to the Internal Diseases (Internal Medicine) outpatient clinic of Necmettin Erbakan University Meram Medical Faculty Hospital, who are at the same age as the case group, and who have not been diagnosed with any disease by the doctor, and who are willing to participate in the study. Healthy individuals will be interviewed once. The obtained data will be compared with the preoperative data of breast cancer patients.
  Interventions: Other: 3-Day Food Intake Record

INTERVENTIONS:
Other: 3-Day Food Intake Record — Collecting clinical and socio-demographic information, nutritional status, food consumption (dietary intake of advanced glycation end products, dietary total antioxidant capacity, dietary inflammatory index), anthropometric measurements (body weight, height, body composition, handgrip strength, upper-middle arm circumference, waist circumference, hip circumference, triceps skinfold thickness), quality of life, biochemical biomarkers (serum carboxymethyl lysine, advanced glycation end products receptor, the soluble receptor of advanced glycation end products, TNF-α, IL-1β, IL-6, malondialdehyde, 2,4-dinitrophenyl hydrazine, 8-hydroxy-2'-deoxyguanosine, total antioxidant capacity)
  Other Names: Anthropometric Measurements; Serum Advanced Glycation End Products Biomarkers

SUMMARY:
Breast cancer is among the most common types of cancer in the world. Factors such as age, reproduction, nutrition, hormonal, and lifestyle factors also play a role in the etiology of breast cancer. Nutrition can affect cancer metabolism at stages such as carcinogen metabolism, cell, and host defense, cell differentiation, and tumor growth. When investigating nutrition and breast cancer risk, it is important to evaluate the preparation and cooking processes applied to foods. Advanced glycation end products (AGE) are formed as a result of heat treatment applied to foods. There are studies showing that AGEs increase inflammation and oxidative stress in the organism. It is aimed to compare the dietary AGE intake and serum levels of AGE participants with breast cancer and healthy participants and to examine the relationship with serum inflammatory, oxidative stress, DNA damage, and total antioxidant capacity. Patients with breast cancer will be evaluated before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy. The amount the dietary AGE intake, serum markers, nutritional status, and changes in quality of life will be determined.

DETAILED DESCRIPTION:
The Location of the Research: The research is carried out in Konya Necmettin Erbakan University Meram Faculty of Medicine General Surgery, Medical Oncology, and Biochemistry Departments. After obtaining the permission of the ethics committee, official permission was obtained from Necmettin Erbakan University Meram Medical Faculty Hospital Chief Physician to conduct the study.

The Sample Size of the Study: It was calculated by in G * Power 3.1.9.2 the computer program. It was determined by taking into account the mean and standard deviation of the blood advanced glycation end products level variable of previous (3.3 ± 1.2 × 105 arbitrary units (AU) in breast cancer patients, 2.3 ± 0.7 × 105 AU in healthy individuals). Considering that the number of samples in the control and breast cancer groups would be equal, it was determined that both groups should consist of at least 27 individuals with an error margin of d = 1.02, α = 0.05, and a power of 0.95. Considering that there will be losses in the sample, at least 32 individuals will be included in both groups. In this study, all of the patients participating in the research are informed in detail and informed consent forms are obtained from all participants.

Statistical analysis: The data will be assessed using the SPSS 22 statistical software package. Mean, standard deviation, minimum and maximum values of the quantitative data will be calculated, and the number and percentage tables of the qualitative data will be created.

In the comparison of quantitative data of the case group (before surgery) and control group, the Student t-test will be used for the normal distribution, and the Mann-Whitney U test will be used for the non-normal distribution. The chi-squared test will be used to evaluate qualitative data.

In the comparison of quantitative data of the case group during follow-up (before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy) one-way ANOVA will be used for the normal distribution, and the Friedman test will be used for the non-normal distribution.

While determining the correlation between quantitative data, the Pearson correlation coefficient will be used for normal distribution and the Spearman correlation coefficient will be used for non-normal distribution.

The p-value < 0.05 was considered to be statistically significant at the end of the analysis.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of breast cancer for the first time, Non-metastatic, Written informed consent

Exclusion Criteria:

Age < 19 years and > 64 years, Metastatic, Pregnancy, Lactation, Clinical diagnosis of moderate/severe neurological impairment, Clinical diagnosis of moderate/severe cognitive impairment, Clinical diagnosis of type 1 diabetes mellitus, Clinical diagnosis of type 2 diabetes mellitus, Refusal to participate

Ages: 19 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Breast cancer occurs almost entirely in female.
Study Population: Case group: The study will include female individuals aged 19-64 years who applied to Necmettin Erbakan University Meram Medical Faculty General Surgery and Medical Oncology Departments and were diagnosed with breast cancer for the first time and volunteering to participate in the study.
  Control group: The control group consists of healthy adult women who applied to the Internal Diseases (Internal Medicine) outpatient clinic of Necmettin Erbakan University Meram Medical Faculty Hospital, who are at the same age as the case group, and who have not been diagnosed with any disease by the doctor, and who are willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Dietary Advanced Glycation End Products Intake (kilounit/day) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  The amount of dietary carboxy methyl lysine intake is calculated using daily food consumption. Previous studies will be used for the carboxy methyl lysine content of foods.
Serum carboxy methyl lysine (CML) level (pg/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It will be determined with ELISA.
Serum receptor for advanced glycation end products (RAGE) level (pg/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It will be determined with ELISA.
Serum soluable receptor for advanced glycation end products (sRAGE) level (pg/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It will be determined with ELISA.
Serum tumor necrosis factor alfa (TNF-α) level (pg/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  Tumor necrosis factor alfa (TNF-α) will be determined with ELISA.
Serum interleukin 1 beta (IL-1β) level (pg/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  Interleukin 1 beta (IL-1β) will be determined with ELISA.
Serum interleukin 6 (IL-6) level (pg/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  Interleukin 6 (IL-6) will be determined with ELISA.
Serum lipid peroxidation level: Malondialdehyde (nmol/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  Malondialdehyde will be determined with ELISA.
Serum protein oxidation level:2,4-Dinitrophenylhydrazine (nmol/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  2,4-Dinitrophenylhydrazine will be determined with ELISA.
Serum DNA damage level: 8-hydroxy 2 deoxyguanosine(ng/mL) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  8-hydroxy 2 deoxyguanosine will be determined with ELISA.
Serum total antioxidant capacity (μmol/L) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It will be determined with spectrophotometric assay.
Dietary total antioxidant capacity: Total Oxygen Radical Absorbans Capacity (T-ORAC) (µmol Trolox equivalent) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It is calculated by using tables published in previous articles.
Dietary total antioxidant capacity: Lipophilic Oxygen Radical Absorption Capacity (L-ORAC)(µmol Trolox equivalent) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It is calculated by using tables published in previous articles.
Dietary total antioxidant capacity: Hydrophilic Oxygen Radical Absorption Capacity (L-ORAC)(µmol Trolox equivalent) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It is calculated by using tables published in previous articles.
Dietary total antioxidant capacity:Trolox Equivalent Antioxidant Capacity (TEAC) (mmol Trolox equivalent) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It is calculated by using tables published in previous articles.
Dietary total antioxidant capacity:Total Radical Trapping Antioxidant Parameter (TRAP) (mmol Trolox equivalent) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It is calculated by using tables published in previous articles.
Dietary total antioxidant capacity:Ferric Reducing Antioxidant Potential (FRAP)(mmol) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  It is calculated by using tables published in previous articles.
Dietary inflammatory index (score) | 15 months (Case group:before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy, For control group: When healthy participant comes to the internal medicine clinic for a routine examination)
  The inflammatory load value will be calculated by using energy, carbohydrate, protein, total fat, cholesterol, saturated fatty acids, monounsaturated fatty acids, polyunsaturated fatty acids, n-3 and n-6 polyunsaturated fatty acids, vitamins (vitamin B12, B9, B6, B3, B2, B1, A, C, D and E) micronutrients (iron, zinc, selenium, magnesium), caffeine, tea, garlic, onion, pepper and β-carotene intake. The resulting value for each dietary factor was multiplied by the inflammatory score of each item to achieve the dietary factor dietary inflammatory index score. Then, all dietary factor dietary inflammatory index scores were summed to calculate the DII score for each participant.
Nutritional status | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  The malnutrition status and severity of participants with breast cancer are determined with Patient Generated Subjective Global Assessment (PG-SGA) test.

SECONDARY OUTCOMES:
Body weight (kg) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  Body weight is measured in lightly dressed clothing without shoes by using an electronic scale sensitive to 100 g.
Height (cm) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  Height is measured using stadiometer in the position of Frankfort plane without shoes.
Body mass index (kg/m2) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  Body mass index (BMI) is calculated by dividing body weight in kilograms by height in metres squared.
Body composition (%) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  The percentages of body fat, body water and lean body mass are measured through bioelectrical impedance analysis.
Handgrip strength (kg) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  Handgrip strength is measured using a handgrip dynamometer.
Mid-upper arm circumference (cm) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  Mid-Upper Arm Circumference (MUAC) is the circumference of the left upper arm, measured at the mid-point between the tip of the shoulder and the tip of the elbow (olecranon process and the acromium).
Triceps skinfold thickness (mm) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  The triceps skinfold is measured at the back of the left arm, midway between the acromial process of the scapula and the olecranon process of the ulna.
Waist circumference (cm | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  Waist circumference is measured at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest
Hip circumference (cm) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  Hip circumference is measured around the widest portion of the buttocks.
Quality of life score-Case group (European Cancer Research and Treatment Organization Quality of Life Scale - Cancer 30 (EORTC QLQ-C30) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  The quality of life of women with breast cancer is evaluated with the European Cancer Research and Treatment Organization Quality of Life Scale - Cancer 30 (EORTC QLQ-C30). It consists of 30 items to assess physical, role, emotional, cognitive and social functioning, global health status or qualitiy of life scales, fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties. Items are measured using a 4-point Likert Scale ranging from Not at all (1) to Very much (4). The lowest score obtained from the scale is 0, the highest score is 100. Higher scores represent higher general health and functional scores and higher scores indicate higher symptom severity.
Quality of life score-Case group (the European Cancer Research and Treatment Organization Breast Cancer-Specific Quality of Life Scale ) | 15 months (Before surgery, before chemotherapy, and in the sixth and twelfth months after starting chemotherapy)
  The EORTC QLQ-BR23 is a breast-specific module that comprises of 23 questions to assess body image, sexual functioning, sexual enjoyment, future perspective, systemic therapy side effects, breast symptoms, arm symptoms and upset by hair loss. Items measured using 4-point Likert Scale ranging from Not at all (1) to Very much (4). The lowest score obtained from the scale is 0, the highest score is 100. Higher scores represent higher functional scores and higher scores indicate higher symptom severity.
Quality of life score-Control group (Short-Form 36-Item Health Survey ) | 3 months
  Short-Form 36-Item Health Survey questionnaire is used to determine the quality of life levels of healthy women.The questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). A final item, termed self-reported health transition, is answered by the client but is not included in the scoring process. The SF-36 offers a choice of recall format at a standard (4 week) or acute (1 week) time frame. Likert scales and yes/no options are used to assess function and well-being on this 36-item questionnaire. Obtained score ranges from 0 to 100. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

REFERENCES:
- [Background] Alpar R. Spor, sağlık ve eğitim bilimlerinden örneklerle uygulamalı istatistik ve geçerlik-güvenirlik. Ankara: Detay Yayıncılık; 2016.
- [Background] Tesarova P, Kalousova M, Jachymova M, Mestek O, Petruzelka L, Zima T. Receptor for advanced glycation end products (RAGE)--soluble form (sRAGE) and gene polymorphisms in patients with breast cancer. Cancer Invest. 2007 Dec;25(8):720-5. doi: 10.1080/07357900701560521. PMID 18058469
- [Background] Shivappa N, Hebert JR, Rosato V, Montella M, Serraino D, La Vecchia C. Association between the dietary inflammatory index and breast cancer in a large Italian case-control study. Mol Nutr Food Res. 2017 Mar;61(3):10.1002/mnfr.201600500. doi: 10.1002/mnfr.201600500. Epub 2016 Nov 30. PMID 27794170
- [Background] Bauer J, Capra S, Ferguson M. Use of the scored Patient-Generated Subjective Global Assessment (PG-SGA) as a nutrition assessment tool in patients with cancer. Eur J Clin Nutr. 2002 Aug;56(8):779-85. doi: 10.1038/sj.ejcn.1601412. PMID 12122555
- [Background] Carlsen MH, Halvorsen BL, Holte K, Bohn SK, Dragland S, Sampson L, Willey C, Senoo H, Umezono Y, Sanada C, Barikmo I, Berhe N, Willett WC, Phillips KM, Jacobs DR Jr, Blomhoff R. The total antioxidant content of more than 3100 foods, beverages, spices, herbs and supplements used worldwide. Nutr J. 2010 Jan 22;9:3. doi: 10.1186/1475-2891-9-3. PMID 20096093
- [Background] Demiral Y, Ergor G, Unal B, Semin S, Akvardar Y, Kivircik B, Alptekin K. Normative data and discriminative properties of short form 36 (SF-36) in Turkish urban population. BMC Public Health. 2006 Oct 9;6:247. doi: 10.1186/1471-2458-6-247. PMID 17029646
- [Background] Demirci S, Eser E, Ozsaran Z, Tankisi D, Aras AB, Ozaydemir G, Anacak Y. Validation of the Turkish versions of EORTC QLQ-C30 and BR23 modules in breast cancer patients. Asian Pac J Cancer Prev. 2011;12(5):1283-7. PMID 21875283
- [Background] Halvorsen BL, Carlsen MH, Phillips KM, Bohn SK, Holte K, Jacobs DR Jr, Blomhoff R. Content of redox-active compounds (ie, antioxidants) in foods consumed in the United States. Am J Clin Nutr. 2006 Jul;84(1):95-135. doi: 10.1093/ajcn/84.1.95. PMID 16825686
- [Background] Pellegrini N, Serafini M, Colombi B, Del Rio D, Salvatore S, Bianchi M, Brighenti F. Total antioxidant capacity of plant foods, beverages and oils consumed in Italy assessed by three different in vitro assays. J Nutr. 2003 Sep;133(9):2812-9. doi: 10.1093/jn/133.9.2812. PMID 12949370
- [Background] Pellegrini N, Serafini M, Salvatore S, Del Rio D, Bianchi M, Brighenti F. Total antioxidant capacity of spices, dried fruits, nuts, pulses, cereals and sweets consumed in Italy assessed by three different in vitro assays. Mol Nutr Food Res. 2006 Nov;50(11):1030-8. doi: 10.1002/mnfr.200600067. PMID 17039458
- [Background] Uribarri J, Woodruff S, Goodman S, Cai W, Chen X, Pyzik R, Yong A, Striker GE, Vlassara H. Advanced glycation end products in foods and a practical guide to their reduction in the diet. J Am Diet Assoc. 2010 Jun;110(6):911-16.e12. doi: 10.1016/j.jada.2010.03.018. PMID 20497781
- [Background] Wu X, Beecher GR, Holden JM, Haytowitz DB, Gebhardt SE, Prior RL. Lipophilic and hydrophilic antioxidant capacities of common foods in the United States. J Agric Food Chem. 2004 Jun 16;52(12):4026-37. doi: 10.1021/jf049696w. PMID 15186133
- [Background] Wu X, Gu L, Holden J, Haytowitz DB, Gebhardt SE, Beecher G, Prior RL. Development of a database for total antioxidant capacity in foods: a preliminary study. Journal of Food Composition and Analysis.2004; 17(3): 407-422.
- [Background] Zujko ME, Witkowska AM. Antioxidant Potential and Polyphenol Content of Selected Food. International Journal of Food Properties.2011; 14(2): 300-308.
- [Background] Zujko ME, Witkowska AM. Antioxidant Potential and Polyphenol Content of Beverages, Chocolates, Nuts, and Seeds. International Journal of Food Properties. 2014; 17(1): 86-92.